CLINICAL TRIAL: NCT07101913
Title: Incidence and Risk Factors of Acute Kidney Injury (AKI) After Anti-CD19 CAR-T Cells Treatments in B-cell Lymphoma and Long Term Evolution.
Brief Title: Occurrence of Acute Kidney Injury After CAR-T Cells Treatments in B-cell Lymphoma.
Acronym: AKI CAR
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5297
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Acute Kidney Injury (AKI); Infusion of CD19 CAR T Cell; B Cell Lymphoma
Keywords: Acute kidney injury/ CD19 CAR T cells
MeSH Terms: conditions — Acute Kidney Injury; Lymphoma, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- CAR-T cells treatment: All patients followed in haematology center in "Hospices civils de Lyon" for a B-cell lymphoma and treated by anti-CD19 CAR-T cells.
  Interventions: Biological: Incidence of acute kidney injury; Other: Describe risk factors in AKI occurrence.; Other: Focus on patient with chronic kidney disease at baseline; Other: Long term evolution after treatment by CAR-T cells

INTERVENTIONS:
Biological: Incidence of acute kidney injury — * Creatinine measurement before lymphodepletion chemotherapy, before CAR-T cells injection (day 0) and at day 1, day 3, day 5, day 7, day 10, day 14, day 21 and day 28.
  * AKI according to 2012 KDIGO.
Other: Describe risk factors in AKI occurrence. — Comparison of caracteristics between participants with AKI and participants without AKI :
  * Baseline caracteristics of participants : age, gender, BMI (Body mass index), medical history…
  * Caracteristics of hematology disease : severity of lymphoma, previous treatments (chemotherapy, autologous/allogenic stem cell transplant), type of CAR-T cells (axi-cel, tisa-cel)
  * Other adverse affects : cytokine release syndrome (CRS), immune effector cell-associated neurotoxicity syndrome (ICANS)
  * Use of nephrotoxic medications Informations found in medical field.
Other: Focus on patient with chronic kidney disease at baseline — Looking at the subgroup with chronic kidney disease at baseline : are the outcomes different in this population ? Efficacity of CAR-T ? More adverse effects ?
Other: Long term evolution after treatment by CAR-T cells — Creatinine measurement 1 year after CAR-T treatment. Informations found in medical field.

SUMMARY:
The investigators want to describe the incidence of AKI after CAR-T cells therapy in B-cell lymphoma. With the aim of highlight risk factors in AKI occurrence. Then, look at outcomes in the subgroup with chronic kidney disease at baseline. Finally, the investigators will examine long term evolution of kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed in haematology center in "Hospices civils de Lyon"
* For a B-cell lymphoma
* Treated by anti-CD19 CAR-T cells

Exclusion Criteria:

* Less than 18 years old
* Patients with legal protection measure
* CAR-T cells therapy for another disease : leukemia, autoimmune disease…

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients followed in haematology center in "Hospices civils de Lyon" for a B-cell lymphoma and treated by anti-CD19 CAR-T cells.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of AKI after CAR-T cell therapy in B-cell lymphoma. In percentage, according to the 2012 KDIGO. | AKI from the day of the injection of CAR-T cells, until 28 days after the injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology department, Centre hospitalier Lyon Sud, Pierre-Bénite, France, France